CLINICAL TRIAL: NCT01049984
Title: A Double-blind, Placebo Controlled, Randomized, Multicenter Study to Assess the Safety and Clinical Benefit of Rasagiline as an Add on Therapy to Stable Dose of Dopamine Agonists in the Treatment of Early Parkinson's Disease
Brief Title: Rasagiline as Add on to Dopamine Agonists in the Treatment of Parkinson's Disease
Acronym: ANDANTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TVP-1012/PM103
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; UPDRS; Clinical Global Evaluation Illness Severity score; Clinical Global Evaluation Improvement; B-SIT; SCOPA - Sleep Daytime Sleepiness; PDQ -39; SCOPA - Cognition; Levodopa; rasagiline; Dopamine Agonist Therapy; monoamine oxidase type B inhibitor
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline 1 mg (Experimental): Participants took a 1 mg rasagiline tablet orally each day for 18 weeks.
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): Participants took a matching placebo tablet once daily for 18 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — 1mg tablet daily for 18 weeks
  Other Names: TVP-1012; AZILECT®
  Arms: Rasagiline 1 mg
Drug: Placebo — one tablet daily for 18 weeks
  Arms: Placebo

SUMMARY:
To assess the efficacy of rasagiline 1 mg as a first add-on treatment to dopamine agonist therapy in early Parkinson Disease (PD) patients, , not optimally controlled on dopamine agonists as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* receiving stable dose of oral ropinirole or pramipexole whose symptoms are not optimally controlled or whose oral dopamine agonist titration regimen was truncated due to intolerability:
* 1) Minimum dose of agonist will be 6 mg/day for ropinirole and 1.0 mg/day for pramipexole
* 2) Stable dopamine agonist treatment must have been ongoing for ≥ 30 days, no longer than 5 years preceding baseline
* Males and females. Women of childbearing potential must agree to practice an acceptable method of birth control.
* Idiopathic Parkinson Disease confirmed at baseline by presence of at least 2 cardinal signs (resting tremor, bradykinesia, rigidity), w/o other known or suspected cause of Parkinsonism
* Hoehn & Yahr > 1 (symptoms on only one side of the body) with treatment and < 3 (mild to moderate bilateral disease; some postural instability; physically independent).
* Dopamine agonist dose must be stable for ≥30 days preceding the baseline visit.
* For patients who are receiving amantadine or anticholinergics, the dose must have been stable for ≥30 days prior to screening.
* Medically stable outpatients (Investigator's judgment).

Exclusion Criteria:

* receive rasagiline or other monoamine oxidase (MAO) inhibitors 60 days preceding baseline
* receive levodopa > 21 consecutive days within 90 days prior baseline
* moderate to severe motor fluctuations
* hepatic impairment
* investigational medications 30 days preceding baseline
* dopamine agonist use > 5 years prior to baseline
* major depression as defined by Beck Depression Inventory (BDI) short form score greater than 14
* significant cognitive impairment as defined by Mini-Mental State Exam (MMSE) score less than 26.
* impulse control disorder (ICD) based on the Questionnaire for Impulsive-compulsive Disorders in Parkinson's Disease form (QUIP).
* pregnant or lactating or planning on becoming pregnant in the next 18 weeks
* uncontrolled hypertension. Patients whose hypertension is controlled with medications are eligible.
* Concomitant monoamine oxidase (MAO) inhibitors or medicines contraindicated w/ MAO inhibitors not allowed

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azhar Choudhry, M.D., Study Director — Teva Neuroscience, Inc.
Locations (58):
- United States (58):
  - Teva Investigational Site 34, Phoenix, Arizona
  - Teva Investigational Site 42, Sun City, Arizona
  - Teva Investigational Site 15, Fountain Valley, California
  - Teva Investigational Site 19, Fresno, California
  - Teva Investigational Site 36, Fresno, California
  - Teva Investigational Site 04, La Jolla, California
  - Teva Investigational Site 29, Reseda, California
  - Teva Investigational Site 69, San Francisco, California
  - Teva Investigational Site 02, Sunnyvale, California
  - Teva Investigational Site 43, Ventura, California
  - Teva Investigational Site 44, Fairfield, Connecticut
  - Teva Investigational Site 07, Manchester, Connecticut
  - Teva Investigational Site 25, Newark, Delaware
  - Teva Investigative Site 63, Atlantis, Florida
  - Teva Investigational Site 30, Boca Raton, Florida
  - Teva Investigational Site 13, Clearwater, Florida
  - Teva Investigational Site 70, Sunrise, Florida
  - Teva Investigational Site 41, Tampa, Florida
  - Teva Investigational Site 61, Vero Beach, Florida
  - Teva Investigational Site 01, Decatur, Georgia
  - Teva Investigational Site 58, Boise, Idaho
  - Teva Investigational Site 49, Glenview, Illinois
  - Teva Investigational Site 23, Peoria, Illinois
  - Teva Investigational Site 47, Indianapolis, Indiana
  - Teva Investigational Site 67, Indianapolis, Indiana
  - Teva Investigational Site 76, Indianapolis, Indiana
  - Teva Investigational Site 55, Des Moines, Iowa
  - Teva Investigational Site 17, Lexington, Kentucky
  - Teva Investigational Site 27, Paducah, Kentucky
  - Teva Investigational Site 56, Scarborough, Maine
  - Teva Investigational Site 62, Elkridge, Maryland
  - Teva Investigational Site 51, Springfield, Massachusetts
  - Teva Investigational Site 11, Detroit, Michigan
  - Teva Investigational Site 33, West Bloomfield, Michigan
  - Teva Investigational Site 39, Golden Valley, Minnesota
  - Teva Investigational Site 22, St Louis, Missouri
  - Teva Investigational Site 08, Great Falls, Montana
  - Teva Investigational Site 59, Missoula, Montana
  - Teva Investigational Site 60, Las Vegas, Nevada
  - Teva Investigational Site 14, Somerset, New Jersey
  - Teva Investigational Site 03, Commack, New York
  - Teva Investigational Site 38, Plainview, New York
  - Teva Investigational Site 05, Asheville, North Carolina
  - Teva Investigational Site 31, Charlotte, North Carolina
  - Teva Investigational Site 28, Raleigh, North Carolina
  - Teva Investigational Site 26, Fargo, North Dakota
  - Teva Investigational Site 35, Cincinnati, Ohio
  - Teva Investigational Site 68, Cincinnati, Ohio
  - Teva Investigational Site 64, Tulsa, Oklahoma
  - Teva Investigational Site 21, Medford, Oregon
  - Teva Investigational Site 40, Portland, Oregon
  - Teva Investigative Site 65, Cordova, Tennessee
  - Teva Investigational Site 71, Brownwood, Texas
  - Teva Investigational Site 18, San Antonio, Texas
  - Teva Investigational Site 32, Temple, Texas
  - Teva Investigational Site 09, Richmond, Virginia
  - Teva Investigational Site 46, Virginia Beach, Virginia
  - Teva Investigational Site 77, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rasagiline 1 mg | Placebo
Started | 163 | 165
Safety Population | 162 (One patient was randomized but not dosed; omitted from safety population) | 164 (One patient was randomized but not dosed; omitted from safety population)
Modified Intent-to-treat Pop | 159 (Took >= 1 dose of study drug and had both baseline and at least 1 post-baseline efficacy assessment) | 162 (Took >= 1 dose of study drug and had both baseline and at least 1 post-baseline efficacy assessment)
Completed | 144 | 146
Not Completed | 19 | 19
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Protocol Violation | 3 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 13 | 7
Not completed — Treatment failure | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasagiline 1 mg | Placebo | Total
Number analyzed (Participants) | 162 | 164 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.27) | 62.8 (10.06) | 62.5 (9.67)
Age, Customized [Number; unit: participants]
  30 to <65 years | 97 | 89 | 186
  65 to <75 years | 49 | 60 | 109
  >=75 years | 16 | 15 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 109 | 111 | 220
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 154 | 155 | 309
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 3 | 7 | 10
  White | 156 | 151 | 307
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Parkinson's Disease Duration [Mean (Standard Deviation); unit: years] — Years since first diagnosis. Data based on the modified intent to treat population of 159, 162 participants.
  years | 2.19 (2.224) | 2.07 (1.940) | 2.13 (2.083)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 18 in the Unified Parkinson's Disease Rating Scale (UPDRS) Total Score for Parts I, II and III
Description: The UPDRS was developed as a comprehensive tool to monitor the impact of Parkinson's Disease and the degree of disability caused. Version 3 of UPDRS contains four parts, three of which are totaled and reported in this outcome. Part I is a clinician's evaluation of mentation (mental activity or state of mind), cognition (ability to acquire knowledge), behaviour and mood. Part II is the participants' evaluation of the disease's impact on normal activities. Part III is a clinician's evaluation of motor function. Parts I, II, and III contain a total of 31 questions, which are each rated on a scale of 0 (normal or no disease effect) to 4 (maximum negative effect), for a total scale of 0-124. Negative change from baseline values indicate improvement.
  All site raters (medical doctor [MD], doctor of osteopathy [DO], nurse practitioner, or physician assistant) received training on how to complete the UPDRS. The same site rater completed the UPDRS at all visits.
Time Frame: Day 0 (baseline), Week 18
Population: Modified intent to treat population - all randomized participants who took at least 1 dose of study drug and had both a baseline and at least 1 post-baseline efficacy assessment. Several participants had missing UPDRS items at baseline and during treatment; therefore the total UPDRS for these participants was set as missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1 mg | Placebo
Number analyzed (Participants) | 158 | 157
units on a scale | -3.6 (0.68) | -1.2 (0.68)
Statistical Analysis 1: Comparison: Rasagiline 1 mg vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA — All analyses were performed at the 2-sided 0.05 significance level. P values were not adjusted; Repeated measures model with baseline score as a covariate and factors Treatment, Week in Study, Pooled Center and Week by Treatment interaction; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.3 to -0.5]

2. Secondary Outcome: Change From Baseline to Week 18 in the Unified Parkinson's Disease Rating Scale (UPDRS) Total Score for Part II - Activities of Daily Living
Description: The UPDRS was developed as a comprehensive tool to monitor the impact of Parkinson's Disease and the degree of disability caused. UPDRS contains four parts, the second of which is reported in this outcome. Part II is the participants' evaluation of the disease's impact on normal activities. Part II contains a total of 13 questions, which are each rated on a scale of 0 (normal or no disease effect) to 4 (maximum negative effect), for a total scale of 0-52. Negative change from baseline values indicate improvement.
Time Frame: Day 0 (baseline), Week 18
Population: Modified intent to treat population - all randomized participants who took at least 1 dose of study drug and had both a baseline and at least 1 post-baseline efficacy assessment. Several participants had missing UPDRS items at baseline and during treatment for subscale II, and therefore that subscale was set as missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1 mg | Placebo
Number analyzed (Participants) | 158 | 160
units on a scale | -0.1 (0.27) | 0.3 (0.27)
Statistical Analysis 1: Comparison: Rasagiline 1 mg vs Placebo; Test type: Superiority or Other; p = 0.301, ANCOVA — All analyses were performed at the 2-sided 0.05 significance level. P values were not adjusted; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.3]

3. Secondary Outcome: Change From Baseline to Week 18 in the Unified Parkinson's Disease Rating Scale (UPDRS) Total Score for Part III - Motor Function
Description: The UPDRS was developed as a comprehensive tool to monitor the impact of Parkinson's Disease and the degree of disability caused. Version 3 of UPDRS contains four parts, the third of which is reported in this outcome. Part III is a clinician's evaluation of motor function. Part III contains 14 questions, which are each rated on a scale of 0 (normal or no disease effect) to 4 (maximum negative effect), for a total scale of 0-56. Negative change from baseline values indicate improvement.
  All site raters (medical doctor [MD], doctor of osteopathy [DO], nurse practitioner, or physician assistant) received training on how to complete the UPDRS. The same site rater completed the UPDRS at all visits
Time Frame: Day 0 (baseline), Week 18
Population: Modified intent to treat population - all randomized participants who took at least 1 dose of study drug and had both a baseline and at least 1 post-baseline efficacy assessment. Several participants had missing UPDRS items at baseline and during treatment for subscale III, and therefore that subscale was set as missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline 1 mg | Placebo
Number analyzed (Participants) | 159 | 158
units on a scale | -3.4 (0.48) | -1.6 (0.48)
Statistical Analysis 1: Comparison: Rasagiline 1 mg vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — All analyses were performed at the 2-sided 0.05 significance level. P values were not adjusted; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.1 to -0.5]

4. Secondary Outcome: Clinical Global Improvement (CGI) Score at Week 18 As Assessed by the Site Rater
Description: CGI is used by the site rater to rate participants total improvement during the study whether or not, in the investigators' judgment, it is due entirely to drug treatment. Specifically, site raters are asked to compare the participants condition at the beginning of the study to his/her condition at Week 18, how much has he/she changed? Answers are 0 (not assessed), 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), 7(very much worse).
  Site raters can be the medical doctor [MD], doctor of osteopathy [DO], nurse practitioner, or physician assistant.
Time Frame: 18 weeks
Population: Modified intent to treat
Measure: Number; unit: participants
Arm/Group | Rasagiline 1 mg | Placebo
Number analyzed (Participants) | 159 | 162
participants
  Not assessed (0) | 0 | 1
  Very much improved (1) | 5 | 5
  Much improved (2) | 21 | 20
  Minimally improved (3) | 45 | 39
  No change (4) | 63 | 53
  Minimally worse (5) | 21 | 42
  Much worse (6) | 3 | 1
  Very much worse (7) | 1 | 1
Statistical Analysis 1: Comparison: Rasagiline 1 mg vs Placebo; Test type: Superiority or Other; p = 0.255, Cochran-Mantel-Haenszel — All analyses were performed at the 2-sided 0.05 significance level. P values were not adjusted. Only participants with assessment (>0) are included in the CMH test; CMH used the proportion of participants in each category between the two treatment arms, with treatment and pooled center as strata

5. Secondary Outcome: Clinical Global Improvement (CGI) Score at Week 18 As Assessed by the Participant
Description: CGI is used by the participant to rate his/her total improvement during the study. Specifically, participants are asked to compare their condition at the beginning of the study to his/her condition at Week 18, how much has he/she changed? Answers are 0 (not assessed), 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), 7(very much worse).
Time Frame: 18 weeks
Population: Modified intent to treat
Measure: Number; unit: participants
Arm/Group | Rasagiline 1 mg | Placebo
Number analyzed (Participants) | 159 | 162
participants
  Not assessed (0) | 0 | 1
  Very much improved (1) | 7 | 7
  Much improved (2) | 18 | 18
  Minimally improved (3) | 39 | 40
  No change (4) | 52 | 52
  Minimally worse (5) | 36 | 35
  Much worse (6) | 5 | 8
  Very much worse (7) | 2 | 1
Statistical Analysis 1: Comparison: Rasagiline 1 mg vs Placebo; Test type: Superiority or Other; p = 0.996, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]

6. Secondary Outcome: Illness Severity Score at Day 0 and Week 18 As Assessed by the Site Rater
Description: Site raters were asked: Considering your total clinical experience with the particular population, how ill is the patient at this time? Answers were based on a 0-7 scale, with 0=not assessed, 1= normal, not at all ill, and 7= among the most extremely ill of patients.
  Site raters can be the medical doctor [MD], doctor of osteopathy [DO], nurse practitioner, or physician assistant.
Time Frame: Day 0 (baseline), Week 18
Population: Modified intent to treat
Measure: Number; unit: participants
Arm/Group | Rasagiline 1 mg | Placebo
Number analyzed (Participants) | 159 | 162
participants
  Day 0: Not assessed (0) | 0 | 0
  Day 0: Normal, not at all ill (1) | 4 | 5
  Day 0: Borderline ill (2) | 18 | 26
  Day 0: Mildly Ill (3) | 95 | 100
  Day 0: Moderately Ill (4) | 39 | 28
  Day 0: Markedly ill (5) | 1 | 2
  Day 0: Severely ill (6) | 0 | 0
  Day 0: Among the most extremely ill (7) | 0 | 0
  Week 18: Not assessed (0) | 0 | 2
  Week 18: Normal, not at all ill (1) | 10 | 5
  Week 18: Borderline ill (2) | 28 | 33
  Week 18: Mildly ill (3) | 90 | 89
  Week 18: Moderately ill (4) | 29 | 31
  Week 18: Markedly ill (5) | 2 | 1
  Week 18: Severely ill (6) | 0 | 1
  Week 18: Among the most extremely ill (7) | 0 | 0
Statistical Analysis 1: Comparison: Rasagiline 1 mg vs Placebo; Test type: Superiority or Other; p = 0.967, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; CMH used the proportion of participants in each category between the two treatment arms, with treatment, pooled center, and baseline value as strata

ADVERSE EVENTS:
Time Frame: Day 0 (post treatment) to Week 18
Arm/Group | Placebo | Rasagiline 1 mg
Serious Adverse Events (participants affected / at risk) | 5/164 | 8/162
Other Adverse Events (participants affected / at risk) | 44/164 | 55/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=164) | Rasagiline 1 mg (N=162)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=164) | Rasagiline 1 mg (N=162)
NAUSEA (Gastrointestinal disorders) | 7 (7) | 10 (10)
OEDEMA PERIPHERAL (General disorders) | 7 (8) | 12 (12)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 9 (9)
DIZZINESS (Nervous system disorders) | 10 (11) | 12 (14)
HEADACHE (Nervous system disorders) | 7 (8) | 10 (15)
SOMNOLENCE (Nervous system disorders) | 11 (11) | 11 (11)
TREMOR (Nervous system disorders) | 10 (10) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. Sponsor may remove information that is considered confidential and/or proprietary other than Study data and results.